CLINICAL TRIAL: NCT03525639
Title: Cardiac Magnetic Resonance Evaluation of Myocardial Inflammation Persistence After Acute Myocarditis: Prognostic Relevance
Brief Title: CMR Evaluation of Myocardial Inflammation Persistence After Acute Myocarditis: Prognostic Relevance
Acronym: MIAMI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Antonio Esposito (Other)
Collaborators: Ministry of Health, Italy (Other Government)
Responsible Party: Sponsor-Investigator, Antonio Esposito, Professor, IRCCS San Raffaele
Organization: IRCCS San Raffaele (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MIAMI GR-2013-02356832
Record Dates: First submitted 2018-05-03; First posted 2018-05-15 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2021-04

CONDITIONS: Myocarditis Acute; Myocardial Inflammation
Keywords: Cardiac Magnetic Resonance; Acute Myocarditis; Myocardial Inflammation
MeSH Terms: conditions — Myocarditis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Acute Myocarditis (Experimental): Patients undergoing Cardiac Magnetic Resonance at baseline, 2 month, 1 year.
  Interventions: Diagnostic Test: Cardiac Magnetic Resonance

INTERVENTIONS:
Diagnostic Test: Cardiac Magnetic Resonance — Additional CMR study 2 month after the initial diagnosis of acute myocarditis to assess myocardial inflammation persistence (2-month-CMR).

SUMMARY:
Patients with acute myocarditis (AM) usually experience spontaneous healing, but a considerable percentage of them evolve towards chronic long-term cardiac impairment. The evolution towards dilated cardiomyopathy (DCM) occurs in a subtle manner, frequently after an initial recover that mimics complete healing. Differences in the course of the disease may reflect the course of underlying myocardial inflammation related to viral clearance or persistence and to the following autoimmune response.

Cardiac magnetic resonance (CMR) mapping parameters have been developed for the quantification of edema and necrosis, showing high diagnostic accuracy. No mapping parameter has been developed for the assessment of the third Lake Louise criteria, namely the hyperemia, and, furthermore, their prognostic role is not completely understood.

The study hypothesis is that the early-enhanced T1 mapping parameter may have great diagnostic accuracy for myocarditis, and that a short-term monitoring with a complete CMR protocol at 2 month after symptoms onset may identify the subgroup of patients at high risk of progression towards DCM.

The results of this study will help to significantly improve diagnostic performances of CMR and may help to manage patients with AM.

DETAILED DESCRIPTION:
Background and Significance:

In patients with acute myocarditis (AM), spontaneous improvement can be observed in the majority of cases, but progression towards dilated cardiomyopathy (DCM) is a not rare outcome (around 20% of patients) (Feldmann N Engl J Med 2000;343:1388-98). Differences in the course of the disease may reflect the course of the underlying viral infection. In a large series of patients with AM submitted to two endo-myocardial biopsies (EMBs) in few months, Kuhl demonstrated that viral clearance was associated with spontaneous ejection fraction (EF) improvement, while EF did not improve or even deteriorated in patients with viral and myocardial inflammation persistence (Kühl Circulation 2005;111:887-93. Kühl Circulation 2005;112:1965-70). However, repeated EMBs cannot be proposed in the clinical routine and, hence, non-invasive detection of the subgroup of patients with inflammation persistence should have important implications. Today, cardiac magnetic resonance (CMR) is recognized as an accurate non-invasive imaging tool to diagnose acute myocarditis, because of its ability to detect myocardial inflammation and necrosis (Friedrich J Am Coll Cardiol 2009;53:1475-87).

The introduction of mapping techniques has significantly improved CMR sensitivity, allowing to detect both focal and diffuse involvement, with a substantial benefit in the convalescent phase where conventional Lake Louise criteria often fail.

However, no technical development has been performed for the evaluation of Early Gadolinium Enhancement (EGE), which continues to be assessed on T1-w images, being the less robust Lake Louise criteria and eliminated from the updated Lake Louise criteria [Ferreira J Am Coll Cardiol 2018;72(24):3158-76.].

Therefore, there are two major clinical needs: (a) the first being the improvement in diagnosis fulfilling the lack in technical advancement in the setting of EGE evaluation, (b) the second being risk-stratification and prediction of prognosis. The study hypothesis is that the development of a quantitative method based on T1 mapping for the assessment of EGE may be highly sensitive and specific for the diagnosis of myocarditis. Then, the assessment of early changes in CMR parameters at a short-term CMR study (2 months after symptoms onset) may have great value in outcome prediction.

Preliminary data: A previous study performed on patients with chronic inflammatory cardiomyopathy demonstrated that the positivity of CMR parameters of necrosis (LGE) and inflammation (oedema) is significantly higher in patients with an active inflammation at EMB, compared to patients with borderline histological criteria (De Cobelli 2006 JACC;47:1649-54). These data suggest the possibility to detect with CMR the persistence of subtle myocardial inflammation after the acute phase in patients with myocarditis.

Moreover, Wagner and Colleagues demonstrated, in a small group of patients, a correlation between CMR evidence of myocardial hyperaemia persistence 4 weeks after the onset of acute myocarditis and negative left ventricular (LV) remodelling 30 months later (Wagner A 2003 MAGMA;16:17-20).

Materials and Methods:

This is a prospective multicentre cohort study. 80 patients with diagnosis of acute myocarditis (AM) will be enrolled.

All patients admitted to Hospital with suspect of AM will be submitted to:

collection of detailed anamnesis and physical examination, 12-lead ECG, laboratory exams, transthoracic echocardiography, coronary catheterization or coronary computed tomography (CT) angiography when an ischemic cause of symptoms need to be excluded and CMR imaging within 3-5 days.

CMR protocol will include Lake-Louise criteria, parametric mappings (native T1, T2 mapping and ECV), with an additional early-enhanced T1 mapping acquired 2 minutes after gadolinium injection.

All patients with clinically or EMB confirmed diagnosis of AM will be enrolled and will undergo a second CMR study 2 month later.

All patients will undergo a clinical/instrumental follow-up including: CMR assessment of LV ejection fraction and end-diastolic volume after at least 1 year from diagnosis; registration of all-cause mortality, cardiac death and aborted cardiac sudden death in patients with implantable cardioverter-defibrillator (ICD).

Impact and Translational Implications:

Myocarditis is characterized by significant heterogeneity of long-term evolution. CMR could play a key role in the non-invasive and early identification of patients with persistent myocardial inflammation, at high risk to evolve towards an irreversible post-myocarditis heart failure. Thus, CMR may help to design tailored management of patients. In this perspective, invasive characterization of damage mechanism and aetiology might be reserved to patients with CMR evidence of inflammation persistence.

ELIGIBILITY:
Inclusion Criteria:

* Presence of at least 1 of the subsequent clinical features [12]:

  * Acute chest pain (pericarditic, or pseudo-ischaemic)
  * New-onset dyspnoea at rest or during exercise
  * Fatigue with or without left/right heart failure signs
  * Palpitation or unexplained arrhythmia symptoms or syncope or aborted sudden cardiac death
  * Unexplained cardiogenic shock
* Associated with at least 1 of the subsequent diagnostic criteria [12]:

  * Newly abnormal 12 lead ECG and/or Holter and/or stress testing, any of the following: I to III degree atrioventricular block, or bundle branch block, ST/T wave change, sinus arrest, ventricular tachycardia or fibrillation and asystole, atrial fibrillation, reduced R wave height, intraventricular conduction delay, abnormal Q waves, low voltage, frequent premature beats, supraventricular tachycardia
  * Myocardial injury markers (elevated troponin T/Troponin I)
  * New, otherwise unexplained left ventricular (LV) and/or right ventricular (RV) functional and/or structural abnormalities on cardiac imaging (echo/angio/CMR) compatible with acute myocarditis and excluding other diseases
* Signed informed consent

Exclusion Criteria:

* History of cardiomyopathies
* Coronary artery disease (coronary catheterization or CT angiography will be performed when coronary artery disease need to be excluded in consideration of signs and symptoms)
* ICD or pacemaker
* Inability to hold breath or to lay down for 45 min
* Claustrophobia
* Recent history of alimentary/alcoholic/respiratory intoxication
* CMR diagnostic criteria suggestive of other cardiac disease explaining signs and symptoms (e.g. myocardial infarction with patent coronary arteries, tako-tsubo syndrome)
* Risk for nephrogenic systemic fibrosis (estimated glomerular filtration rate < 30 mL/min/1.73 m2)
* History of allergic reaction to MR contrast media
* Pregnancy or breast-feeding

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-12-06 (Actual); Primary Completion 2020-12-31 (Actual); Study Completion 2021-02-20 (Actual)

PRIMARY OUTCOMES:
Improvement in CMR diagnosis with early enhanced T1 mapping and early changes in CMR parameters reflecting inflammation activity | Baseline; 2 month
  T2 ratio; LGE (Late Gadolinium Enhancement); native T1 relaxation time; T2 relaxation time; extracellular volume fraction (ECV); early enhanced T1 relaxation time; baseline; 2 month; delta (2 month - baseline).
MACE and left ventricular remodelling | Inclusion; 2 month
  Major adverse cardiac events (MACE): cardiac death; aborted sudden cardiac death; all-cause mortality.
  Left ventricular end-diastolic volume (LV EDV); left ventricular ejection fraction (LVEF).

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Esposito, Principal Investigator — IRCCS San Raffaele
Locations (3):
- Italy (3):
  - IRCCS San Raffaele, Milan
  - Policlinico Umberto I, Roma
  - AOU Città della Salute e della Scienza, Torino

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Youn JC, Shim HS, Lee JS, Ji AY, Oh J, Hong N, Lee HS, Park S, Lee SH, Choi D, Chung N, Kang SM. Detailed pathologic evaluation on endomyocardial biopsy provides long-term prognostic information in patients with acute myocarditis. Cardiovasc Pathol. 2014 May-Jun;23(3):139-44. doi: 10.1016/j.carpath.2014.01.004. Epub 2014 Jan 17. PMID 24529879
- [Background] Anzini M, Merlo M, Sabbadini G, Barbati G, Finocchiaro G, Pinamonti B, Salvi A, Perkan A, Di Lenarda A, Bussani R, Bartunek J, Sinagra G. Long-term evolution and prognostic stratification of biopsy-proven active myocarditis. Circulation. 2013 Nov 26;128(22):2384-94. doi: 10.1161/CIRCULATIONAHA.113.003092. Epub 2013 Oct 1. PMID 24084750
- [Background] Sagar S, Liu PP, Cooper LT Jr. Myocarditis. Lancet. 2012 Feb 25;379(9817):738-47. doi: 10.1016/S0140-6736(11)60648-X. Epub 2011 Dec 18. PMID 22185868
- [Background] Kuhl U, Pauschinger M, Noutsias M, Seeberg B, Bock T, Lassner D, Poller W, Kandolf R, Schultheiss HP. High prevalence of viral genomes and multiple viral infections in the myocardium of adults with "idiopathic" left ventricular dysfunction. Circulation. 2005 Feb 22;111(7):887-93. doi: 10.1161/01.CIR.0000155616.07901.35. Epub 2005 Feb 7. PMID 15699250
- [Background] Kuhl U, Pauschinger M, Seeberg B, Lassner D, Noutsias M, Poller W, Schultheiss HP. Viral persistence in the myocardium is associated with progressive cardiac dysfunction. Circulation. 2005 Sep 27;112(13):1965-70. doi: 10.1161/CIRCULATIONAHA.105.548156. Epub 2005 Sep 19. PMID 16172268
- [Background] Friedrich MG, Sechtem U, Schulz-Menger J, Holmvang G, Alakija P, Cooper LT, White JA, Abdel-Aty H, Gutberlet M, Prasad S, Aletras A, Laissy JP, Paterson I, Filipchuk NG, Kumar A, Pauschinger M, Liu P; International Consensus Group on Cardiovascular Magnetic Resonance in Myocarditis. Cardiovascular magnetic resonance in myocarditis: A JACC White Paper. J Am Coll Cardiol. 2009 Apr 28;53(17):1475-87. doi: 10.1016/j.jacc.2009.02.007. PMID 19389557
- [Background] Mahrholdt H, Wagner A, Deluigi CC, Kispert E, Hager S, Meinhardt G, Vogelsberg H, Fritz P, Dippon J, Bock CT, Klingel K, Kandolf R, Sechtem U. Presentation, patterns of myocardial damage, and clinical course of viral myocarditis. Circulation. 2006 Oct 10;114(15):1581-90. doi: 10.1161/CIRCULATIONAHA.105.606509. Epub 2006 Oct 2. PMID 17015795
- [Background] Natale L, De Vita A, Baldari C, Meduri A, Pieroni M, Lombardo A, Crea F, Bonomo L. Correlation between clinical presentation and delayed-enhancement MRI pattern in myocarditis. Radiol Med. 2012 Dec;117(8):1309-19. doi: 10.1007/s11547-012-0790-x. Epub 2012 Feb 10. English, Italian. PMID 22327917
- [Background] Grun S, Schumm J, Greulich S, Wagner A, Schneider S, Bruder O, Kispert EM, Hill S, Ong P, Klingel K, Kandolf R, Sechtem U, Mahrholdt H. Long-term follow-up of biopsy-proven viral myocarditis: predictors of mortality and incomplete recovery. J Am Coll Cardiol. 2012 May 1;59(18):1604-15. doi: 10.1016/j.jacc.2012.01.007. Epub 2012 Feb 22. PMID 22365425
- [Background] Caforio AL, Pankuweit S, Arbustini E, Basso C, Gimeno-Blanes J, Felix SB, Fu M, Helio T, Heymans S, Jahns R, Klingel K, Linhart A, Maisch B, McKenna W, Mogensen J, Pinto YM, Ristic A, Schultheiss HP, Seggewiss H, Tavazzi L, Thiene G, Yilmaz A, Charron P, Elliott PM; European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Current state of knowledge on aetiology, diagnosis, management, and therapy of myocarditis: a position statement of the European Society of Cardiology Working Group on Myocardial and Pericardial Diseases. Eur Heart J. 2013 Sep;34(33):2636-48, 2648a-2648d. doi: 10.1093/eurheartj/eht210. Epub 2013 Jul 3. PMID 23824828
- [Background] De Cobelli F, Pieroni M, Esposito A, Chimenti C, Belloni E, Mellone R, Canu T, Perseghin G, Gaudio C, Maseri A, Frustaci A, Del Maschio A. Delayed gadolinium-enhanced cardiac magnetic resonance in patients with chronic myocarditis presenting with heart failure or recurrent arrhythmias. J Am Coll Cardiol. 2006 Apr 18;47(8):1649-54. doi: 10.1016/j.jacc.2005.11.067. Epub 2006 Mar 29. PMID 16631005
- [Background] Wagner A, Schulz-Menger J, Dietz R, Friedrich MG. Long-term follow-up of patients paragraph sign with acute myocarditis by magnetic paragraph sign resonance imaging. MAGMA. 2003 Feb;16(1):17-20. doi: 10.1007/s10334-003-0007-7. PMID 12695882
- [Background] Francone M, Chimenti C, Galea N, Scopelliti F, Verardo R, Galea R, Carbone I, Catalano C, Fedele F, Frustaci A. CMR sensitivity varies with clinical presentation and extent of cell necrosis in biopsy-proven acute myocarditis. JACC Cardiovasc Imaging. 2014 Mar;7(3):254-63. doi: 10.1016/j.jcmg.2013.10.011. Epub 2014 Feb 19. PMID 24560214
- [Background] Frustaci A, Russo MA, Chimenti C. Randomized study on the efficacy of immunosuppressive therapy in patients with virus-negative inflammatory cardiomyopathy: the TIMIC study. Eur Heart J. 2009 Aug;30(16):1995-2002. doi: 10.1093/eurheartj/ehp249. Epub 2009 Jun 25. PMID 19556262
- [Background] Chimenti C, Kajstura J, Torella D, Urbanek K, Heleniak H, Colussi C, Di Meglio F, Nadal-Ginard B, Frustaci A, Leri A, Maseri A, Anversa P. Senescence and death of primitive cells and myocytes lead to premature cardiac aging and heart failure. Circ Res. 2003 Oct 3;93(7):604-13. doi: 10.1161/01.RES.0000093985.76901.AF. Epub 2003 Sep 4. PMID 12958145
- [Background] Yeon SB, Salton CJ, Gona P, Chuang ML, Blease SJ, Han Y, Tsao CW, Danias PG, Levy D, O'Donnell CJ, Manning WJ. Impact of age, sex, and indexation method on MR left ventricular reference values in the Framingham Heart Study offspring cohort. J Magn Reson Imaging. 2015 Apr;41(4):1038-45. doi: 10.1002/jmri.24649. Epub 2014 May 12. PMID 24817313
- [Background] Luetkens JA, Doerner J, Thomas DK, Dabir D, Gieseke J, Sprinkart AM, Fimmers R, Stehning C, Homsi R, Schwab JO, Schild H, Naehle CP. Acute myocarditis: multiparametric cardiac MR imaging. Radiology. 2014 Nov;273(2):383-92. doi: 10.1148/radiol.14132540. Epub 2014 Jun 6. PMID 24910904
- [Background] Mason JW. Myocarditis and dilated cardiomyopathy: an inflammatory link. Cardiovasc Res. 2003 Oct 15;60(1):5-10. doi: 10.1016/s0008-6363(03)00437-1. PMID 14522402
- [Background] Kuhl U, Pauschinger M, Schwimmbeck PL, Seeberg B, Lober C, Noutsias M, Poller W, Schultheiss HP. Interferon-beta treatment eliminates cardiotropic viruses and improves left ventricular function in patients with myocardial persistence of viral genomes and left ventricular dysfunction. Circulation. 2003 Jun 10;107(22):2793-8. doi: 10.1161/01.CIR.0000072766.67150.51. Epub 2003 May 27. PMID 12771005
- [Background] Frustaci A, Chimenti C, Calabrese F, Pieroni M, Thiene G, Maseri A. Immunosuppressive therapy for active lymphocytic myocarditis: virological and immunologic profile of responders versus nonresponders. Circulation. 2003 Feb 18;107(6):857-63. doi: 10.1161/01.cir.0000048147.15962.31. PMID 12591756
- [Background] Ferreira VM, Schulz-Menger J, Holmvang G, Kramer CM, Carbone I, Sechtem U, Kindermann I, Gutberlet M, Cooper LT, Liu P, Friedrich MG. Cardiovascular Magnetic Resonance in Nonischemic Myocardial Inflammation: Expert Recommendations. J Am Coll Cardiol. 2018 Dec 18;72(24):3158-3176. doi: 10.1016/j.jacc.2018.09.072. PMID 30545455